CLINICAL TRIAL: NCT00784732
Title: A Randomized, Partially-blinded, Placebo-controlled, Two-way Crossover, Proof of Concept Study to Compare the Relative Efficacy of CRTh2 Receptor Antagonist, QAV680 Against Placebo in the Treatment of Allergic Rhinitis in an Environmental Exposure Chamber (EEC) Model
Brief Title: A Study to Compare the Efficacy of QAV680 Against Placebo in Treating Seasonal Allergic Rhinitis in an Environmental Exposure Chamber
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQAV680A2202
Record Dates: First submitted 2008-11-03; First posted 2008-11-04 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Seasonal Allergic Rhinitis; Environmental Exposure Chamber; nasal lavage
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — NVP-QAV680; Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: QAV680
- 2 (Experimental)
  Interventions: Drug: QAV680
- 3 (Active Comparator)
  Interventions: Drug: Mometasone Furoate

INTERVENTIONS:
Drug: QAV680
  Arms: 1
Drug: QAV680
  Arms: 2
Drug: Mometasone Furoate
  Arms: 3

SUMMARY:
This study will compare the effectiveness of QAV680 against placebo in treating the symptoms of seasonal allergic rhinitis in an Environmental Exposure Chamber.

ELIGIBILITY:
Inclusion Criteria:

* Positive skin prick test to ragweed allergen
* FEV1 must be ≥80% predicted value at screening and prior to entry into EEC on Day -2.
* Patients must weigh at least 50 kg, and must have a body mass index (BMI) within the range of 18 to 35 kg/m2.
* Non-smokers and ex-smokers (≤10 pack years and >6 months of smoking abstinence).
* Understand and sign the written informed consent

Exclusion Criteria:

* Patients requiring a change in the use of any prescription drugs within four (4) weeks prior to initial dosing.
* Participation in any clinical investigation within four (4) weeks prior to initial dosing or longer if required by local regulations, and for any other limitation of participation based on local regulations.
* Significant illness within two (2) weeks prior to initial dosing.
* History of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result.
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Total Nasal Symptom Score (TNSS) over the last 2 hours of exposure in the EEC Percentage nasal lavage eosinophil count post EEC | TNSS: 6-8h during EEC exposure on Day 10

SECONDARY OUTCOMES:
Measure of nasal cytokines (ECP, IL-5, IL-13, PGD2, Eotaxin) | After 8h exposure in EEC
Absolute eosinophil count from nasal lavage collected | During exposure in EEC
Nasal airway patency assessed by acoustic rhinometry during exposure in the EEC | During exposure in EEC
Total Ocular Symptom Score measured during exposure in the EEC | During exposure in EEC
Assess pharmacokinetics of plasma QAV680 in patients with seasonal allergic rhinitis | Through out study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis Investigator Site
Locations (1):
- Novartis Investigator Site, Toronto, Canada